CLINICAL TRIAL: NCT03338738
Title: Impact of Beta-lactams on the Microbiota and Relative Fecal Abundance of Multidrug Resistant Bacteria Ans Its Importance on Infectious Episodes in Hospitalized Patients
Brief Title: Impact of Beta-lactams on the Microbiota and Relative Fecal Abundance of Mulltidrug Resistant Bacteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Hospital Avicenne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COPROBLSE
Record Dates: First submitted 2017-10-19; First posted 2017-11-09 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Enterobacterial Infection
MeSH Terms: conditions — Enterobacteriaceae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with ESBL, antibiotic pressure (Experimental): Patients with ESBL, antibiotic pressure will be included. On the day of inclusion, a stool culture is performed on the first stool issued after the start of antibiotic therapy in order to evaluate the initial flora and the relative initial faecal abundance of multidrug-resistant bacteria. In the absence of stool emission by the patient, a rectal swab will be performed. 72 hours after initiation of antibiotic therapy, a blood sample (5 ml) will be taken to determine plasma concentrations of antibiotics. In addition, a stool sample will be taken at 72 hours after the start of antibiotic therapy, at the end of antibiotic therapy and 60 days after this end to evaluate the change in initial flora and relative faecal abundance of ESBL-producing enterobacteria.
  Interventions: Diagnostic Test: Stool culture ans swab

INTERVENTIONS:
Diagnostic Test: Stool culture ans swab — Patients with ESBL enterobacteria, antibiotic pressure are patients with ESBL positive result diagnosed by stool culture and a rectal swab.
  The intervention correspond to addition of 4 stool samples (or 4 rectal swabs in the absence of stool emission) and a blood sample.

SUMMARY:
The global spread of ESBL-producing enterobacteria (EBLSE) poses a real public health problem. The exposure of patients to antibiotic therapy leads to an increase in resistant bacterial populations within the digestive flora. As a result, the diagnosis of digestive colonization by EBLSE is an event that has become common in hospitalized patients in intensive care / intensive care under high pressure antibiotics. The aim of this work is to study the impact of beta-lactams frequently prescribed on the microbiota and the emergence of multiresistant bacteria in the digestive flora and to evaluate, in colonized patients, the factors associated with the occurrence of an infectious episode. In particular, the impact of the relative fecal abundance of ESBL enterobacteriaceae on the occurrence of this event will be studied.

DETAILED DESCRIPTION:
Among enterobacteria, the production of ESBL is the first cause of multi-resistance. The consequences of multidrug-resistant enterobacterial infections predominantly represented by ESBLs are currently well known, both from the individual point of view (increase in mortality and length of hospital stay) and collective (increase in costs of care). Data from the literature reveal an increased risk of ESBL bacteremia in patients with rectal carriage of ESBL-producing enterobacteria. It therefore appears necessary in known patients with ESBL-producing enterobacteria to evaluate the impact of different antibiotics (beta-lactams) on the modification of flora, the increase of faecal abundance in multidrug-resistant bacteria such as E. coli ESBL and evaluate the factors associated with infections in these patients.

ELIGIBILITY:
Inclusion Criteria:

* age> 18
* ICU admitted patient
* rectal colonization of Enterobacteria
* accepting participation
* with medical insurance

Exclusion Criteria:

* patient without bacterial colonization
* under antibiotics more than 24hours
* without medical insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
percentage of EBLSE | Day 60
  ratio of number of colony of enterobacteria BLSE on number of total bacteria colony

CONTACTS AND LOCATIONS:
Overall Officials: ZAHAR Jean Ralph, Professor, Study Chair — AVICENNE HOSPITAL; LE MONNIER Alban, Professor, Study Director — GHPSJ
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Pilmis B, Mizrahi A, Pean de Ponfilly G, Philippart F, Bruel C, Zahar JR, Le Monnier A. Relative faecal abundance of extended-spectrum beta-lactamase-producing Enterobacterales and its impact on infections among intensive care unit patients: a pilot study. J Hosp Infect. 2021 Jun;112:92-95. doi: 10.1016/j.jhin.2021.03.022. Epub 2021 Mar 29. PMID 33794294